CLINICAL TRIAL: NCT06929156
Title: A Multi-center, Single-dose, Open-label, Parallel Design, Pharmacokinetics Study of BGM0504 Injection in Healthy Participants and Participants With Impaired Renal Function
Brief Title: A Study of BGM0504 in Healthy Participants and Participants With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-I-101
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Overweight or Obese
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- A group (Healthy Control) (Experimental)
  Interventions: Drug: BGM0504
- B group (Mild Renal Impairment) (Experimental)
  Interventions: Drug: BGM0504
- C group (Moderate Renal Impairment) (Experimental)
  Interventions: Drug: BGM0504
- D group (Severe Renal Impairment) (Experimental)
  Interventions: Drug: BGM0504

INTERVENTIONS:
Drug: BGM0504 — Receive a single dose of BGM0504 injection
  Arms: A group (Healthy Control)
Drug: BGM0504 — Receive a single dose of BGM0504 injection
  Arms: B group (Mild Renal Impairment)
Drug: BGM0504 — Receive a single dose of BGM0504 injection
  Arms: C group (Moderate Renal Impairment)
Drug: BGM0504 — Receive a single dose of BGM0504 injection
  Arms: D group (Severe Renal Impairment)

SUMMARY:
The purpose of this study is to assess how fast BGM0504 gets into the blood stream and how long it takes the body to remove it in participants with impaired kidney function compared to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* √ Age 18-65 years on the date of signing informed consent (inclusive);

  * Body mass index (BMI) within the range of 19.0-30.0 kg/m2 (inclusive);.
  * Stable renal function, assessed by two eGFR during screening (apart at least 3 days);
  * Diagnosed as stable, chronic renal disease for at least 3 months.
  * Renal function, assessed by estimated glomerular filtration rate at screening (eGFR):

    1. Normal renal function: 90-129 mL/min (inclusive);
    2. Mild impairment: 60-89 mL/min (inclusive);
    3. Moderate impairment: 30-59 mL/min (inclusive);
    4. Severe impairment: 15-29 mL/min (inclusive);

Exclusion Criteria:

* ● Allergic constitution includes severe drug allergy or history of drug allergy;

  * Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2; Have a history or presence of pancreatitis;
  * Participants in clinical trials of any drug or medical device in the 3 months prior to screening;.
  * Suspected or confirmed history of alcohol or drug abuse;
  * Hepatitis B surface antigen (HBsAg), HIV antibody detection, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
  * Donation or loss of 200 mL or more of blood within 3 months prior to screening, or blood donation during screening or within 1 months after the end of the trial;
  * Pregnant or Breast-feeding women;
  * The investigator considers that the participant has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve (AUC) of BGM0504 From Time Zero to Tlast (AUC0-t) | Start of Treatment up to Day 29
  Area Under the Concentration Versus Time Curve (AUC) of BGM0504 From Time Zero to Tlast (AUC0-t)
Maximum Concentration of BGM0504 (Cmax) | Start of Treatment up to Day 29
  Maximum Concentration of BGM0504 (Cmax)
Area Under the Concentration Versus Time Curve (AUC) of BGM0504 From Time Zero to Infinity (AUC0-inf) | Start of Treatment up to Day 29
  Area Under the Concentration Versus Time Curve (AUC) of BGM0504 From Time Zero to Infinity (AUC0-inf)

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Start of Treatment up to Day 29
  Time to maximum concentration (Tmax)
Apparent terminal half-life (t1/2) | Start of Treatment up to Day 29
  Apparent terminal half-life (t1/2)
Apparent clearance (CL/F) | Start of Treatment up to Day 29
  Apparent clearance (CL/F)
Incidence and severity of adverse events | Screening period up to Day 29
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Qianfoshan Hospital, Shandong Province), Jinan, Shandong, China